CLINICAL TRIAL: NCT05134805
Title: Functional Outcomes of Hemiarthroplasty Versus Cephalo-medullary Fixation in the Treatment of Unstable Intertrochanteric Femoral Fractures
Brief Title: Outcomes of Hemiarthroplasty Versus Cephalo-medullary Fixation to Treat Unstable Intertrochanteric Femoral Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Islam Mohamed Soliman, Orthopaedic surgery specialist- Principal investigator, Amiri Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU M D 308 2018
Record Dates: First submitted 2021-11-13; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Fracture of Femur
Keywords: BHA , PFN , HHS
MeSH Terms: conditions — Femoral Fractures | interventions — Fracture Fixation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BHA group (Other): Patients will undergo Bipolar hemiarthroplasty operation
  Interventions: Procedure: Bipolar hemiarthroplasty , proximal femoral nail
- PFN group (Other): Patients will undergo cehphalo-medullary fixation (Proximal femoral nail)
  Interventions: Procedure: Bipolar hemiarthroplasty , proximal femoral nail

INTERVENTIONS:
Procedure: Bipolar hemiarthroplasty , proximal femoral nail — * Removal of head of femur , greater trochanter , and lesser trochanter and use bioplar hemiarthroplasty (BHA).
  * Intra-medullary fixation of intertrchanteric femoral fracture by proximal femoral nail (PFN) Fixation of the fracture by using intramedullary nail(proximal femoral nail).
  Other Names: prosthetic joint , fracture fixation

SUMMARY:
Comparing functional outcomes of hemiarthroplasty (prosthetic joint) versus cephalo-medullary fixation ( proximal femoral intramedullary nail) in the treatment of unstable intertrochanteric femoral fractures (proximal femur fractures) in elderly people above 60 years old.

DETAILED DESCRIPTION:
The intertrochanteric femoral fractures incidence rate has increased through the last years because of increasing life expectancy, leading to more morbidity and mortality rates . Unstable fracture pattern occurs due to age increase and bone quality decrease. Unstable intertrochanteric femoral fractures (ITFF) are considered about 40-45% of hip fractures in elderly people . Of note, 55% of these fractures had unstable patterns . The main objective of treatment is to restore the patients to their preoperative daily activities and medical conditions .

Therefore, the surgical treatment aims to return the patient to his pre-fracture level of activity to ensure that the patient moves as soon as possible to prevent complications due to immobility which can lead to death.

In an unstable fracture pattern which is characterized by decreased bone quality, it is of great importance to providing efficient and proper treatment . A lot of treatment modalities had been used in the treatment of this fracture pattern such as PFN, unipolar hemiarthroplasty, BHA, and dynamic hip screw (DHS) . On the other hand, it is difficult to perform stable fixation owing to osteoporotic bone quality.

The treatment aims to restore the patient's ambulation and decrease medical complications and technical failure. By using either BHA or PFN methods, patients can return to pre-injury levels decreasing complications induced by prolonged immobilization or implant failure .

The primary objective of the current study is to compare functional outcomes of unstable ITFF managed by PFN or BHA among cases with ages more than 60 years old. The second main objective is to compare intraoperative and postoperative in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 60 years old.
* Unstable intertrochanteric femoral fractures

Exclusion Criteria:

* patient with age less than 60 years old
* Hip osteoarthritis
* Pathological fractures
* Bilateral fractures
* Metabolic bone disease
* Multiple trauma

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
-Harris Hip Score(HHS) | First 3 months post-operative
  - Harris Hip Score(HHS) : scale from 70 to 100 (70-90) . The higher the HHS, the less dysfunction. A total score of <70 is considered a poor result; 70-80 is considered fair, 80-90 is good, and 90-100 is an excellent result (1). No normative values are available.
-Mobility Score (MS) | First 3 months post-operative
  - Mobility score(MS) :
  scale from 0 to 3 (0-3) 0 being good mobility and 3 being severely impaired mobility. The higher mobility score, the higher mobility impairment.

SECONDARY OUTCOMES:
-Harris Hip Score(HHS) | 1 year follow up
  - Harris hip score (HHS):
  scale from 70 to 100 (70-100). The higher the HHS, the less dysfunction. A total score of <70 is considered a poor result; 70-80 is considered fair, 80-90 is good, and 90-100 is an excellent result (1). No normative values are available.
Mobility Score (MS) | 1 year follow up
  - Mobility score(MS) :
  scale from 0 to 3 (0-3) 0 being good mobility and 3 being severely impaired mobility. The higher mobility score, the higher mobility impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed K Asal, MD, Study Director — Ain shams university, Faculty of Medicine
Locations (1):
- Faculty of Medicine, Ain Shams university, Cairo, Abbasia, Egypt

REFERENCES:
- [Background] Emami M, Manafi A, Hashemi B, Nemati A, Safari S. Comparison of intertrochanteric fracture fixation with dynamic hip screw and bipolar hemiarthroplasty techniques. Arch Bone Jt Surg. 2013 Sep;1(1):14-7. Epub 2013 Sep 15. PMID 25207277
- [Background] Lindskog DM, Baumgaertner MR. Unstable intertrochanteric hip fractures in the elderly. J Am Acad Orthop Surg. 2004 May-Jun;12(3):179-90. doi: 10.5435/00124635-200405000-00006. PMID 15161171
- [Background] Blomfeldt R, Tornkvist H, Eriksson K, Soderqvist A, Ponzer S, Tidermark J. A randomised controlled trial comparing bipolar hemiarthroplasty with total hip replacement for displaced intracapsular fractures of the femoral neck in elderly patients. J Bone Joint Surg Br. 2007 Feb;89(2):160-5. doi: 10.1302/0301-620X.89B2.18576. PMID 17322427
- [Background] Roder F, Schwab M, Aleker T, Morike K, Thon KP, Klotz U. Proximal femur fracture in older patients--rehabilitation and clinical outcome. Age Ageing. 2003 Jan;32(1):74-80. doi: 10.1093/ageing/32.1.74. PMID 12540352
- [Background] Gupta KL. COMPARATIVE ASSESSMENT OF PRIMARY AND SECONDARY OUTCOME WITH PFNA AND HEMIARTHROPLASTY FOR SENILE INTERTROCHANTERIC FRACTURES MANAGEMENT: A PROSPECTIVE RANDOMIZED CLINICAL STUDY. International Journal of Medical and Biomedical Studies (IJMBS). 2020;4(3):205-8.
- [Background] Maru N, Rasik D, Parag T. Unstable intertrochanteric fractures in high risk elderly patients treated with primary bipolar hemiarthroplasty: retrospective case series. Int J Orthop. 2019;5:616-9.
- [Background] Harris WH. Traumatic arthritis of the hip after dislocation and acetabular fractures: treatment by mold arthroplasty. An end-result study using a new method of result evaluation. J Bone Joint Surg Am. 1969 Jun;51(4):737-55. No abstract available. PMID 5783851
- [Background] Kokoroghiannis C, Aktselis I, Deligeorgis A, Fragkomichalos E, Papadimas D, Pappadas I. Evolving concepts of stability and intramedullary fixation of intertrochanteric fractures--a review. Injury. 2012 Jun;43(6):686-93. doi: 10.1016/j.injury.2011.05.031. Epub 2011 Jul 14. PMID 21752370
- [Background] Gaumetou E, Zilber S, Hernigou P. Non-simultaneous bilateral hip fracture: epidemiologic study of 241 hip fractures. Orthop Traumatol Surg Res. 2011 Feb;97(1):22-7. doi: 10.1016/j.otsr.2010.07.011. Epub 2011 Jan 15. PMID 21239241
- [Background] Han SK, Lee BY, Kim YS, Choi NY. Usefulness of multi-detector CT in Boyd-Griffin type 2 intertrochanteric fractures with clinical correlation. Skeletal Radiol. 2010 Jun;39(6):543-9. doi: 10.1007/s00256-009-0795-6. Epub 2009 Sep 8. PMID 20405284
- [Background] Setiobudi T, Ng YH, Lim CT, Liang S, Lee K, Das De S. Clinical outcome following treatment of stable and unstable intertrochanteric fractures with dynamic hip screw. Ann Acad Med Singap. 2011 Nov;40(11):482-7. PMID 22206063
- [Background] Li J, Chen JK, Zhou K, Shen B, Ni XM, Chen L. [Application of dynamic hip screw with modified reamer in intertrochanteric fracture in the elderly]. Zhongguo Gu Shang. 2011 May;24(5):362-5. Chinese. PMID 21688528
- [Background] Yang YH, Wang YR, Jiang SD, Jiang LS. Proximal femoral nail antirotation and third-generation Gamma nail: which is a better device for the treatment of intertrochanteric fractures? Singapore Med J. 2013 Aug;54(8):446-50. doi: 10.11622/smedj.2013152. PMID 24005451
- [Background] Haentjens P, Lamraski G. Endoprosthetic replacement of unstable, comminuted intertrochanteric fracture of the femur in the elderly, osteoporotic patient: a review. Disabil Rehabil. 2005 Sep 30-Oct 15;27(18-19):1167-80. doi: 10.1080/09638280500055966. PMID 16278186
- [Background] Zhou S, Liu J, Zhen P, Shen W, Chang Y, Zhang H, Zhu Q, Li X. Proximal femoral nail anti-rotation versus cementless bipolar hemiarthroplasty for unstable femoral intertrochanteric fracture in the elderly: a retrospective study. BMC Musculoskelet Disord. 2019 Oct 29;20(1):500. doi: 10.1186/s12891-019-2793-8. PMID 31664982
- [Background] Gormeli G, Korkmaz MF, Gormeli CA, Adanas C, Karatas T, Simsek SA. Comparison of femur intertrochanteric fracture fixation with hemiarthroplasty and proximal femoral nail systems. Ulus Travma Acil Cerrahi Derg. 2015 Dec;21(6):503-8. doi: 10.5505/tjtes.2015.96166. PMID 27054643
- [Background] Jolly A, Bansal R, More AR, Pagadala MB. Comparison of complications and functional results of unstable intertrochanteric fractures of femur treated with proximal femur nails and cemented hemiarthroplasty. J Clin Orthop Trauma. 2019 Mar-Apr;10(2):296-301. doi: 10.1016/j.jcot.2017.09.015. Epub 2017 Sep 29. PMID 30828197
- [Background] Kesmezacar H, Ogut T, Bilgili MG, Gokay S, Tenekecioglu Y. [Treatment of intertrochanteric femur fractures in elderly patients: internal fixation or hemiarthroplasty]. Acta Orthop Traumatol Turc. 2005;39(4):287-94. Turkish. PMID 16269874
- [Background] Kim SY, Kim YG, Hwang JK. Cementless calcar-replacement hemiarthroplasty compared with intramedullary fixation of unstable intertrochanteric fractures. A prospective, randomized study. J Bone Joint Surg Am. 2005 Oct;87(10):2186-92. doi: 10.2106/JBJS.D.02768. PMID 16203881
- [Background] Luo X, He S, Zeng D, Lin L, Li Q. Proximal femoral nail antirotation versus hemiarthroplasty in the treatment of senile intertrochanteric fractures: Case report. Int J Surg Case Rep. 2017;38:37-42. doi: 10.1016/j.ijscr.2017.04.027. Epub 2017 Jul 11. PMID 28734187
- [Background] Boldin C, Seibert FJ, Fankhauser F, Peicha G, Grechenig W, Szyszkowitz R. The proximal femoral nail (PFN)--a minimal invasive treatment of unstable proximal femoral fractures: a prospective study of 55 patients with a follow-up of 15 months. Acta Orthop Scand. 2003 Feb;74(1):53-8. doi: 10.1080/00016470310013662. PMID 12635794
- [Background] Papasimos S, Koutsojannis CM, Panagopoulos A, Megas P, Lambiris E. A randomised comparison of AMBI, TGN and PFN for treatment of unstable trochanteric fractures. Arch Orthop Trauma Surg. 2005 Sep;125(7):462-8. doi: 10.1007/s00402-005-0021-5. PMID 16059696